CLINICAL TRIAL: NCT00413894
Title: An Open Label Study of the Effect of Intravenous Mircera on Hemoglobin Levels in Anemic Patients With Chronic Kidney Disease Who Are on Dialysis, and Who Have Previously Received Epoetin Alfa or Beta or Darbepoetin Alfa Treatment.
Brief Title: A Study of Intravenous Mircera for the Treatment of Anemia in Dialysis Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20572
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — iv monthly, with starting dose based on previous dose of epoetin alfa or beta or darbepoetin alfa

SUMMARY:
This single arm study will assess the efficacy and safety of intravenous Mircera, administered with pre-filled syringes, for the treatment of anemia in patients with chronic kidney disease who are on dialysis, and who have previously received treatment with epoetin alfa or beta or darbepoetin alfa. Patients will receive monthly intravenous injections of Mircera, with the starting dose derived from the dose of epoetin alfa or beta or darbepoetin they were receiving in the week preceding study start. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia;
* longterm hemodialysis for >=12 weeks before screening;
* baseline Hb between 10 and 13g/dL;
* iv or sc maintenance epoetin alfa or beta or darbepoetin alfa therapy with same dosing interval for >=4 weeks before screening.

Exclusion Criteria:

* acute or chronic bleeding within 8 weeks prior to screening;
* transfusion of red blood cells within 8 weeks prior to screening;
* poorly controlled hypertension necessitating interruption of erythropoetin treatment in previous 6 months;
* previous treatment with Mircera.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (88):
- Germany (88):
  - Aachen
  - Alzey
  - Ansbach
  - Augsburg
  - Bad König
  - Bad Nenndorf
  - Bad Oeynhausen
  - Bad Orb
  - Bayreuth
  - Berlin
  - Bochum
  - Bottrop
  - Bovenden
  - Braunschweig
  - Bremen
  - Coesfeld
  - Cologne
  - Darmstadt
  - Daun
  - Demmin
  - Dessau
  - Dortmund
  - Düsseldorf
  - Erfurt
  - Essen
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Freudenstadt
  - Fulda
  - Fürstenzell
  - Fürth
  - Gelsenkirchen
  - Gerolstein
  - Giessen
  - Göttingen
  - Greifswald
  - Gütersloh
  - Halle
  - Hamburg
  - Hannoversch Münden
  - Harsewinkel
  - Heide
  - Heidelberg
  - Heilbronn
  - Hildesheim
  - Homburg
  - Homburg/saar
  - Idar-Oberstein
  - Jena
  - Karlsruhe
  - Kiel
  - Krefeld
  - Lauterbach
  - Leipzig
  - Lennestadt
  - Ludwigsburg
  - Ludwigshafen
  - Lüdenscheid
  - Marburg
  - Marl
  - Meiningen
  - Memmingen
  - Minden
  - Mönchengladbach
  - München
  - Neuruppin
  - Oberschleißheim
  - Offenbach
  - Offenburg
  - Potsdam
  - Recklinghausen
  - Regensburg
  - Reutlingen
  - Ribnitz-Damgarten
  - Rostock
  - Saarbrücken
  - Schloss Holte-stutenbrock
  - Schwerin
  - Schwetzingen
  - Stralsund
  - Stuttgart
  - Trier
  - Waiblingen
  - Weinheim
  - Wiesbaden
  - Wiesloch
  - Wuppertal
  - Würzburg

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694
- [Derived] Fliser D, Kleophas W, Dellanna F, Winkler RE, Backs W, Kraatz U, Fassbinder W, Wizemann V, Strack G. Evaluation of maintenance of stable haemoglobin levels in haemodialysis patients converting from epoetin or darbepoetin to monthly intravenous C.E.R.A.: the MIRACEL study. Curr Med Res Opin. 2010 May;26(5):1083-9. doi: 10.1185/03007991003666652. PMID 20225992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 661 participants with renal anemia due to chronic kidney disease (CKD) were enrolled; of which, 424 participants were treated with methoxy polyethylene glycol-epoetin beta (C.E.R.A) and are included in results.
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta (C.E.R.A): During screening (Month -2 to -1), participants received their previous ESA (Erythropoiesis Stimulating Agent) (epoetin alfa/beta/delta or darbepoetin alfa) at previously applied dosing scheme. During titration (Month 1-5), participants received C.E.R.A. at a starting dose of 125 or 200 micrograms per month (μg/month) administered once monthly intravenously (IV). Doses were subsequently adjusted by investigator according to participant's hemoglobin (Hb) values. During evaluation (Month 6 to 8), participants received C.E.R.A once monthly administered IV at a dose decided by investigator according to participant's Hb values.
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta (C.E.R.A)
Started | 424
Completed | 344
Not Completed | 80
Not completed — Withdrawal by Subject | 10
Not completed — Administrative Reasons | 1
Not completed — Hb <10 grams/deciliter | 12
Not completed — Adverse Event | 28
Not completed — Protocol Violation | 11
Not completed — Other | 18

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of study medication independent of whether they completed the study or not.
Groups:
- C.E.R.A: During screening (Month -2 to -1), participants received their previous ESA (epoetin alfa/beta/delta or darbepoetin alfa) at previously applied dosing scheme. During titration (Month 1-5), participants received C.E.R.A. at a starting dose of 125 or 200 μg/month administered once monthly IV. Doses were subsequently adjusted by investigator according to participant's hemoglobin values. During evaluation (Month 6 to 8), participants received C.E.R.A once monthly administered IV at a dose decided by investigator according to participant's Hb values.
Arm/Group | C.E.R.A
Number analyzed (Participants) | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 258

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hb Levels Within 11.0-12.5 Grams Per Deciliter (g/dL) During Evaluation Phase
Time Frame: Visits 8 to 10 (Months 6 to 8)
Population: Completer Population (CP) included only participants who completed the study until Visit 10 (Month 8).
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 344
percentage of participants | 31.7

2. Primary Outcome: Percentage of Participants With Hb Levels Within 10.0-13.0 g/dL During Evaluation Phase
Time Frame: Visits 8 to 10 (Months 6 to 8)
Population: CP
Measure: Number; unit: percentage of participants
Groups:
- C.E.R.A: During screening (Month -2 to -1), participants received their previous ESA (epoetin alfa/beta/delta or darbepoetin alfa) at previously applied dosing scheme. During titration (Month 1-5), participants received C.E.R.A. at a starting dose of 125 or 200 μg/month administered once monthly IV. Doses were subsequently adjusted by investigator according to participant's hemoglobin values. During evaluation (Month 6 to 8), participants received methoxy C.E.R.A once monthly administered IV at a dose decided by investigator according to participant's Hb values.
Arm/Group | C.E.R.A
Number analyzed (Participants) | 344
percentage of participants | 75.6

3. Primary Outcome: Percentage of Participants With Hb Levels Within 11.0-12.5 g/dL by Dose Modifications During Evaluation Phase
Description: Dose adjustment included increase or decrease in dose. Percentage of participants with Hb levels within 11.0-12.5 g/dL by dose adjustment categories (with dose adjustment and without dose adjustment) were reported.
Time Frame: Visits 8 to 10 (Months 6 to 8)
Population: CP; number (n) equals (=) number of participants in the specified category
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 344
percentage of participants
  Without Dose Modification (n=178) | 44.9
  With Dose Modification (n=166) | 17.5

4. Primary Outcome: Percentage of Participants With Hemoglobin Levels Within 10.0-13.0 g/dL by Dose Modification During Evaluation Phase
Description: as for outcome 3
Time Frame: Visits 8 to 10 (Months 6 to 8)
Population: CP; n = number of participants in the specified category
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 344
percentage of participants
  Without Dose Modification (n=178) | 88.8
  With Dose Modification (n=166) | 61.5

5. Secondary Outcome: Percentage of Participants With Hb Levels Within 11.0-12.5 g/dL During Screening Phase
Time Frame: Visits 1 to 2 (Months -2 to -1)
Population: ITT Population: All participants having received at least one dose of study medication and having at least one Hb value measurement under C.E.R.A. were included.
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 416
percentage of participants | 36.8

6. Secondary Outcome: Percentage of Participants With Hb Levels Within 10.0-13.0 g/dL During Screening Phase
Time Frame: Visits 1 to 2 (Months -2 to -1)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 416
percentage of participants | 91.6

7. Secondary Outcome: Percentage of Participants With Hb Levels Within 11.0-12.5 g/dL by Dose Modification During Screening Phase
Description: as for outcome 3
Time Frame: Visits 1 to 2 (Months -2 to -1)
Population: ITT Population; n = number of participants in the specified category
Measure: Number; unit: percentage of participants
Groups:
- C.E.R.A: During screening (Month -2 to -1), participants received their previous ESA (epoetin alfa/beta/delta or darbepoetin alfa) at previously applied dosing scheme. During titration (Month 1-5), participants received C.E.R.A. at a starting dose of 125 or 200 μg/month administered once monthly IV. Doses were subsequently adjusted by investigator according to participant's hemoglobin values. During evaluation (Month 6 to 8), participants received C.E.R.A monthly administered IV at a dose decided by investigator according to participant's Hb values.
Arm/Group | C.E.R.A
Number analyzed (Participants) | 416
percentage of participants
  Without Dose Modification (n=288) | 43.4
  With Dose Modification (n=128) | 21.9

8. Secondary Outcome: Percentage of Participants With HbLevels Within 10.0-13.0 g/dL by Dose Modification During Screening Phase
Description: as for outcome 3
Time Frame: Visits 1 to 2 (Months -2 to -1)
Population: ITT Population; n = number of participants in the specified category
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 416
percentage of participants
  Without Dose Modification (n=288) | 93.1
  With Dose Modification (n=128) | 88.3

9. Secondary Outcome: Percentage of Participants With Changes Between Screening and Evaluation Phase With Respect To Hb Levels
Description: Shifts in Hb levels between Screening and Evaluation Phase were classified as follows: Category A: Participants with Hb levels in both Screening and Evaluation Phase within 10-13 g/dL; Category B: Participants who had Hb values within 10-13 g/dL during Screening but shifted outside the range during Evaluation; Category C: Participants who had Hb values outside range during Screening but shifted to stable values (at least within 10 - 13 g/dL) during Evaluation.; Category D: Participants with less than two values available during Evaluation Phase.
  Participants could appear in only 1 category. Participants had to have 2 or 3 values within range (depending on the number of measurements available) to be counted.
Time Frame: Visits 1 to 2 (Months -2 to -1) and Visits 8 to 10 (Months 6 to 8)
Population: ITT Population;
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 416
percentage of participants
  Category A | 59.4
  Category B | 19.5
  Category C | 4.3
  Category D | 14.9

10. Secondary Outcome: Percentage of Participants With Hb Fluctuations Within Evaluation Phase
Description: Hb fluctuation was defined as the deviation from individual mean Hb-value within the study phase (Evaluation Phase) and was categorized as less than or equal to (≤) ±1 g/dL, greater than (>) ±1.0 to ±1.5 g/dL, > ±1.5 to ±2.0 g/dL, and > ±2.0 g/dL. Percentage of participants within these deviation categories were reported for Evaluation Phase of the study.
Time Frame: Visits 8 to 10 (Months 6 to 8)
Population: ITT population
Measure: Number; unit: percentage of participants
Groups:
- C.E.R.A: During screening (Month -2 to -1), participants received their previous ESA (epoetin alfa/beta/delta or darbepoetin alfa) at previously applied dosing scheme. During titration (Month 1-5), participants received C.E.R.A. at a starting dose of 125 or 200 μg/month administered once monthly IV. Doses were subsequently adjusted by investigator according to participant's hemoglobin values. During evaluation (Month 6 to 8), participants received methoxy polyethylene glycol-epoetin beta once monthly administered IV at a dose decided by investigator according to participant's Hb values.
Arm/Group | C.E.R.A
Number analyzed (Participants) | 416
percentage of participants
  ≤ ± 1.0 g/dl | 82.9
  > ± 1.0 to ± 1.5 g/d | 7.9
  > ± 1.5 to ± 2.0 g/dl | 2.9
  > ± 2.0 g/dl | 0.5
  Missing | 5.8

11. Secondary Outcome: Percentage of Participants With Hb Fluctuations Within Screening Phase
Description: Hematology and clinical chemistry were performed partially by a central laboratory as well as by the local laboratories by means of their established methods. Normal ranges and methods as well as quality assurance certificates had to be available to the sponsor prior to the start of the study. Hb fluctuation was defined as the deviation from individual mean Hb-value within the study phase (Screening Phase) and was categorized as ≤ ±1 g/dL, >±1.0 to ±1.5 g/dL, >±1.5 to ±2.0 g/dL, and >±2.0 g/dL. Percentage of participants within these deviation categories are reported for Screening Phase of the study.
Time Frame: Visits 1 to 2 (Months -2 to -1)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 416
percentage of participants
  ≤ ± 1.0 g/dl | 90.6
  > ± 1.0 to ± 1.5 g/dl | 8.7
  > ± 1.5 to ± 2.0 g/dl | 0.7

12. Secondary Outcome: Percentage of Participants Requiring Erythrocyte Transfusions
Time Frame: Visits 1 to 10 (Months -2 to 8)
Population: Safety Population (SAF): All participants who received at least one dose of study medication independent from whether they completed the study or not were included into the safety analysis.
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 424
percentage of participants
  During Screening Phase | 0.7
  During Titration or Evaluation Phase | 5.0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded in the Safety Population from Day 1 of study drug administration until the end of follow-up period (up to 60 days after Visit 10)
Arm/Group | C.E.R.A
Serious Adverse Events (participants affected / at risk) | 174/424
Other Adverse Events (participants affected / at risk) | 173/424
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A (N=424)
Anaemia (Blood and lymphatic system disorders) | 7
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1
Acute Coronary Syndrome (Cardiac disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 1
Angina Pectoris (Cardiac disorders) | 1
Angina Unstable (Cardiac disorders) | 2
Aortic Valve Stenosis (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 2
Mitral Valve Disease (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 1
Goitre (Endocrine disorders) | 1
Hyperparathyroidism Secondary (Endocrine disorders) | 1
Glaucoma (Eye disorders) | 1
Vitreous Haemorrhage (Eye disorders) | 1
Acute Abdomen (Gastrointestinal disorders) | 1
Anal Fistula (Gastrointestinal disorders) | 1
Dental Caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Duodenal Ulcer (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Gastritis Erosive (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Inguinal Hernia (Gastrointestinal disorders) | 2
Intestinal Infarction (Gastrointestinal disorders) | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Tooth Socket Haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Application Site Dermatitis (General disorders) | 1
Cardiac Death (General disorders) | 1
Chest Pain (General disorders) | 1
Drug Withdrawal Syndrome (General disorders) | 1
General Physical Health Deterioration (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pain (General disorders) | 2
Systemic Inflammatory Response Syndrome (General disorders) | 1
Ulcer Haemorrhage (General disorders) | 1
Bile Duct Stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Abscess Jaw (Infections and infestations) | 1
Bronchitis Viral (Infections and infestations) | 1
Catheter Related Infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Gangrene (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis Clostridial (Infections and infestations) | 1
Localised Infection (Infections and infestations) | 3
Paronychia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Respiratory Tract Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Shunt Infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 2
Arteriovenous Fistula Site Haemorrhage (Injury, poisoning and procedural complications) | 1
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 1
Decompression Sickness (Injury, poisoning and procedural complications) | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 2
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Respiratory Fume Inhalation Disorder (Injury, poisoning and procedural complications) | 1
Shunt Aneurysm (Injury, poisoning and procedural complications) | 2
Shunt Blood Flow Excessive (Injury, poisoning and procedural complications) | 1
Shunt Malfunction (Injury, poisoning and procedural complications) | 3
Shunt Occlusion (Injury, poisoning and procedural complications) | 11
Shunt Stenosis (Injury, poisoning and procedural complications) | 2
Shunt Thrombosis (Injury, poisoning and procedural complications) | 7
Vascular Bypass Dysfunction (Injury, poisoning and procedural complications) | 1
Arteriogram Coronary (Investigations) | 1
Blood Pressure Increased (Investigations) | 1
Haemoglobin Decreased (Investigations) | 58
Reticulocyte Count Decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Fluid Overload (Metabolism and nutrition disorders) | 1
Fluid Retention (Metabolism and nutrition disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Facet Joint Syndrome (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix Carcinoma Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Penis Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance Disorder (Nervous system disorders) | 2
Cerebral Ischaemia (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Grand Mal Convulsion (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1
Cardiac Neurosis (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Diabetic Nephropathy (Renal and urinary disorders) | 1
Renal Cyst (Renal and urinary disorders) | 2
Renal Failure (Renal and urinary disorders) | 3
Renal Failure Chronic (Renal and urinary disorders) | 8
Breast Mass (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Coronary Angioplasty (Surgical and medical procedures) | 1
Large Intestine Anastomosis (Surgical and medical procedures) | 1
Aortic Stenosis (Vascular disorders) | 1
Arterial Occlusive Disease (Vascular disorders) | 3
Circulatory Collapse (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Ischaemia (Vascular disorders) | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 5
Shock (Vascular disorders) | 1
Subclavian Steal Syndrome (Vascular disorders) | 1
Varicose Vein (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A (N=424)
Diarrhoea (Gastrointestinal disorders) | 49
Nausea (Gastrointestinal disorders) | 36
Vomiting (Gastrointestinal disorders) | 32
Influenza Like Illness (General disorders) | 21
Nasopharyngitis (Infections and infestations) | 53
Bronchitis (Infections and infestations) | 33
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.